CLINICAL TRIAL: NCT06294548
Title: A Phase Ib/II, Dose Escalation and Dose Expansion Study of Valemetostat Tosylate (DS-3201b) With Atezolizumab and Bevacizumab in Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Study of Valemetostat Tosylate (DS-3201b) With Atezolizumab and Bevacizumab in HCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mehmet Akce, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012272 (UAB 23152)
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1b: Valemetostat + Atezolizumab 1200 mg + Bevacizumab 15 mg/kg (Experimental): In Phase 1b patients will receive valemetostat (DS-3201) orally daily at their assigned dose level, plus atezolizumab 1200 mg intravenously (IV) on day 1, and bevacizumab 15 mg/kg IV on day 1 of each cycle.
  During Phase 1b, a 3+3 dose escalation design will be utilized to define the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) with starting dose of valemetostat 150mg by mouth daily.
  Interventions: Drug: Valemetostat; Drug: Atezolizumab; Drug: Bevacizumab
- Phase II: Valemetostat + Atezolizumab 1200 mg + Bevacizumab 15 mg/kg (Experimental): During Phase II, study participants will receive valemetostat (DS-3201) orally daily at MTD/RP2D, plus atezolizumab 1200 mg intravenously (IV) on day 1, and bevacizumab 15 mg/kg IV on day 1 of each cycle.
  Interventions: Drug: Valemetostat; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Valemetostat — Valemetostat is an inhibitor of the enzymes enhancer of zeste homolog 1 (EZH1) and enhancer of zeste homolog 2 (EZH2).
  Other Names: Valemetostat tosylate; Valemetostat (DS-3201)
Drug: Atezolizumab — Atezolizumab is commercially available. Atezolizumab combined with bevacizumab is approved for frontline treatment of advanced HCC based on IMbrave150 clinical trial. It will be administered as per the package insert and institutional standards.
Drug: Bevacizumab — Bevacizumab is commercially available. Bevacizumab combined with atezolizumab is approved for frontline treatment of advanced HCC based on IMbrave150 clinical trial. It will be administered as per the package insert and institutional standards.

SUMMARY:
This is a phase Ib/II, dose escalation and dose expansion study of valemetostat (DS-3201) with atezolizumab and bevacizumab in patients advanced Hepatocellular carcinoma (HCC) who did not receive prior systemic therapy for advanced HCC.

DETAILED DESCRIPTION:
Patients will be started on valemetostat (DS-3201) with atezolizumab and bevacizumab, restaging scans will be performed every 9 weeks. The treatment will be continued until progressive disease (PD), unacceptable toxicity or consent withdrawal. Paired research biopsies will be performed.

This study will enroll up to approximately 45-patients at UAB. It is estimated 2 patients will be enrolled per month over up to 36 months period.

Patients will receive valemetostat (DS-3201) orally daily at their assigned dose level, plus atezolizumab 1200 mg intravenously (IV) on day 1, and bevacizumab 15 mg/kg IV on day 1 of each cycle. Each cycle is 21 days. Atezolizumab and bevacizumab will be administered based on institutional guidelines and practice at the FDA approved dosages and intervals for advanced HCC. Valemetostat should be taken immediately prior to the start of atezolizumab and bevacizumab infusion on day 1 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be eligible for enrollment into the study:

1. Sign and date the informed consent form (ICF), prior to the start of any study-specific qualification procedures.
2. Subjects ≥18 years of age or the minimum legal adult age (whichever is greater) at the time the ICF is signed
3. HCC diagnosis confirmed by histology/cytology or clinically by American Association for Study of Liver Diseases (AASLD) 36 criteria in cirrhotic patients.
4. At least one measurable untreated lesion per RECIST v1.1 (see Section 12). Patients who received prior liver directed therapy (ie., Trans arterial chemoembolization [TACE], Y-90, liver directed radiation etc.) are eligible provided the target lesion(s) have not been previously treated with liver directed therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST v1.1 (See Section 12)
5. Locally advanced, metastatic, or unresectable disease.
6. No prior systemic therapy for advanced HCC.
7. Child Pugh Class A.
8. Barcelona Clinic Liver Cancer (BCLC) Stage B (not amenable to liver directed therapy) or Stage C.
9. ECOG Performance Status (PS) 0 or 1.
10. The following laboratory values obtained ≤ 28 days prior to registration. Local laboratory data must meet the following criteria at both Screening and prior to dosing on the planned Cycle 1 Day 1 visit to confirm relatively preserved organ function:

    * Absolute neutrophil count (ANC) ≥1500/mm3
    * Platelet count 100,000/mm3 (platelet transfusion is not allowed within 14 days prior to screening assessment).
    * Hemoglobin (Hgb) 9.0 g/dL (red blood cell transfusion is not allowed within 14 days prior to screening assessment).
    * Total bilirubin (TBIL) ≤1.5 x ULN.
    * ALT and AST ≤3 x ULN
    * For patients not receiving therapeutic anticoagulation INR or aPTT ≤2 x ULN
    * Creatinine clearance ≥40 mL/min (measured by the Cockcroft-Gault equation)
11. If the subject is a female of childbearing potential, she must have a negative serum pregnancy test at Screening and must be willing to use highly effective birth control, as detailed in Section 4.4, upon enrollment, during the Treatment Period, and for 6 months, following the last dose of study drug. A female is considered of childbearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (undergone a hysterectomy, bilateral salpingectomy or bilateral oophorectomy) with surgery at least 1 month before the first dose of study drug or confirmed by follicle stimulating hormone (FSH) test >40 mIU/mL and estradiol <40 pg/mL (<140 pmol/L).

    If male with partner of childbearing potential, the subject must be surgically sterile or willing to use highly effective birth control (Section 4.4) upon enrollment, during the Treatment Period, and for 6 months following the last dose of study drug.

    Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 6months after the final study drug administration.

    Male subjects must not freeze or donate sperm starting at Screening and throughout the study period, and for at least 6 months after the final study drug administration.
12. Provide informed written consent ≤28 days prior to registration.
13. Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).

    Note: During the Active Monitoring Phase of a study (i.e., active treatment), participants must be willing to return to the consenting institution for follow-up.
14. Willing to provide mandatory blood specimens for correlative research purposes (see Section 10).
15. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE v 5.0, Grade ≤1 or Baseline.

Note: Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to > Grade 2 for at least 3 months prior to enrollment and managed with standard of care treatment), which the Investigator deems related to previous anticancer therapy, composed of the following:

1. Chemotherapy-induced neuropathy.
2. Fatigue.
3. Residual toxicities from prior immunotherapy treatment: Grade 1 or 2 endocrinopathies, which may include the following:

   * Hypothyroidism/ hyperthyroidism.
   * Type I diabetes.
   * Hyperglycemia.
   * Adrenal insufficiency.
   * Adrenalitis.
   * Skin hypopigmentation (vitiligo).

Exclusion Criteria:

Subjects who meet any of the following criteria will be disqualified from entering the study:

1. Any of the following because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

   * Pregnant persons
   * Nursing persons
   * Persons of childbearing potential who are unwilling to employ adequate contraception
2. Liver directed therapy (Trans arterial chemoembolization [TACE], Y-90, liver directed radiation, etc.) ≤ 28 days prior to registration.
3. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
4. Uncontrolled or significant cardiovascular disease, including the following:

   * Evidence of prolongation of QT/QTc interval (eg, repeated episodes of QT corrected for heart rate using Fridericia's method [QTcF] >470 ms) (average of triplicate determinations)
   * Myocardial infarction within 6 months prior to Screening
   * Uncontrolled angina pectoris within 6 months prior to Screening
   * New York Heart Association (NYHA) Class 3 or 4 congestive heart failure
   * Inadequately controlled hypertension (defined as systolic blood pressure ≥150 mmHg and/or diastolic blood pressure >100 mmHg, based on average ≥3 blood pressure readings on ≥2 sessions. Anti-hypertensive therapy to achieve these parameters is allowed.
5. Prior malignancy active within the previous 3 years except for locally curable cancer that is currently considered as cured, such as cutaneous basal or squamous cell carcinoma, superficial bladder cancer, or cervical carcinoma in situ, or an incidental histological finding of prostate cancer.
6. History of treatment with other EZH inhibitors
7. Current use of moderate or strong cytochrome P450 (CYP)3A inducers, and strong CYP3A and/or P-gp inhibitors in dose escalation phase (See Table 11).
8. Immunocompromised patients and patients known to be Human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy or known acquired immunodeficiency syndrome.
9. Regarding hepatitis B, patients must meet the following criteria to be eligible:

   1. Patients with Hepatitis B (positive HBs antigen test) have an HBV-DNA Viral Load <2000 IU/mL off treatment or on oral antiviral therapy for at least 4 weeks and during the participation in the study.
   2. For patients at high-risk of Hepatitis B reactivation: Patients with contact to the Hepatitis B virus (positive HBc antibody) that did not develop immunity (negative HBs antibody) must have an HBV-DNA Viral Load <100 IU/mL on oral antiviral therapy for at least 4 weeks and during the participation in the study.
10. Patient has active Hepatitis C. Active Hepatitis C is defined by a positive Hep C Ab result and quantitative HCV RNA results greater than the lower limits of detection of the assay.
11. Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection requiring treatment with intravenous antibiotics, antivirals, or antifungals. Note: Subjects with localized fungal infections of skin or nails are eligible.
12. A medical history or complication considered inappropriate for participation in the study, or a serious physical or psychiatric disease, the risk of which may be increased by participation in the study in the investigator's opinion.
13. Psychological, social, familial, or geographical factors or substance abuse that would prevent regular follow-up to be compliant with the protocol.
14. History of hemoptysis (≥2.5 mL of bright red blood per episode) within 1 month prior to initiation of study treatment
15. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
16. Current or recent (within 10 days of first dose of study treatment) use of aspirin (> 325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.
17. Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose. Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR < 1.5 x ULN and aPTT is within normal limits within 14 days prior to initiation of study treatment. Prophylactic use of low molecular-weight heparin (i.e., enoxaparin 40 mg/day) is allowed.
18. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to the first dose of bevacizumab.
19. History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment
20. History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding within 6 months prior to initiation of study treatment. Patients with signs/symptoms of sub-/occlusive syndrome/intestinal obstruction at time of initial diagnosis may be enrolled if they had received definitive (surgical) treatment for symptom resolution.
21. Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure.
22. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
23. Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses (< 30 mm from the carina) of large volume Patients with vascular invasion of the portal or hepatic veins may be enrolled.
24. History of intra-abdominal inflammatory process within 6 months prior to initiation of study treatment, including but not limited to peptic ulcer disease, diverticulitis, or colitis
25. Radiotherapy within 28 days and abdominal/ pelvic radiotherapy within 60 days prior to initiation of study treatment, except palliative radiotherapy to bone lesions within 7 days prior to initiation of study treatment
26. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment, or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to initiation of study treatment or anticipation of need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure
27. Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID). Occasional use of NSAIDs for the symptomatic relief of medical conditions such as headache or fever is allowed.
28. Known fibrolamellar carcinoma (FLC), sarcomatoid HCC, or combined hepatocellular-cholangiocarcinoma (cHCC-CC)
29. Patients with untreated or incompletely treated varices with bleeding or high-risk for bleeding. Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months of prior to initiation of study treatment do not need to repeat the procedure.
30. History of allogenic organ transplantation.
31. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
32. History of leptomeningeal carcinomatosis or intracranial metastases
33. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
34. Current or prior use of immunosuppressive medication ≤ 14 days prior to registration. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
35. Receipt of live attenuated vaccine ≤30 days prior to registration. Note: Patients, if enrolled, should not receive live vaccine whilst on study treatment and up to 30 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-08-28 (Estimated)

PRIMARY OUTCOMES:
Phase 1b | Baseline up to 36 months
  Evaluate the safety, tolerability, and MTD/RP2D of valemetostat when administered with atezolizumab and bevacizumab in advanced HCC (phase 1b).
Phase II | Baseline up to 36 months
  Estimate the objective response rate (ORR) by RECIST version 1.1. per investigator assessment for valemetostat when administered with atezolizumab and bevacizumab at RP2D in advanced HCC (phase II).

SECONDARY OUTCOMES:
Safety and pharmacokinetics (PK) | Baseline up to 36 months
  Evaluate the safety and pharmacokinetic (PK) profile of valemetostat in combination with atezolizumab and bevacizumab.
Progression free survival (PFS) | Baseline until the date of objective disease progression or death.
  Estimate progression free survival (PFS) for valemetostat when administered with atezolizumab and bevacizumab in advanced HCC.
Overall survival (OS) | Baseline up to 48 months
  Estimate overall survival (OS) for valemetostat when administered with atezolizumab and bevacizumab in advanced HCC.
Duration of response (DoR) | Baseline up to 48 months
  Estimate duration of response (DoR) for valemetostat when administered with atezolizumab and bevacizumab in advanced HCC.
Disease Control Rate (DCR) | Baseline up to 48 months
  Estimate the disease control rate (DCR) for valemetostat when administered with atezolizumab and bevacizumab in advanced HCC.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akce, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States